CLINICAL TRIAL: NCT03724773
Title: Outcomes of Long-Arm Casting Versus Sugar-Tong Splinting of Displaced Forearm Shaft Fractures
Brief Title: Long-Arm vs Sugar-Tong
Acronym: LAST
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Decided not to enroll
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201807196
Record Dates: First submitted 2018-10-22; First posted 2018-10-30 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Closed Fracture of Shaft of Ulna; Closed Fracture of Shaft of Radius
Keywords: Closed Reduction; Sugar-Tong Splint; Long-Arm Cast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Long-Arm Cast (Active Comparator): Reduction and long-arm cast application will be performed by PGY-1 and up residents with adequate training and/or supervision in the required techniques.
  Interventions: Device: Long-Arm Cast
- Sugar-Tong Splint (Active Comparator): Reduction and sugar-tong splint application will be performed by PGY-1 and up residents with adequate training and/or supervision in the required techniques.
  Interventions: Device: Sugar-Tong Splint

INTERVENTIONS:
Device: Long-Arm Cast — A long-arm cast is a circumferential wrapping of the arm from the fingers to above the elbow with casting material.
  Arms: Long-Arm Cast
Device: Sugar-Tong Splint — A sugar-tong splint is the application of hard splinting material on the front and back of the arm.
  Arms: Sugar-Tong Splint

SUMMARY:
The purpose of this study is to determine whether a sugar-tong splint is as effective as a long-arm cast in maintaining reduction of pediatric forearm shaft fractures in a randomized, prospective manner. Consented participants will be randomly assigned to be treated with either a sugar-tong splint or a long-arm cast (both standard of care treatments) in REDCap. Each participant will have a 50/50 chance of being assign to either treatment.

DETAILED DESCRIPTION:
Forearm fractures are very common in the pediatric population and can often be treated with closed reduction and immobilization. Immobilization techniques include long-arm casting, short-arm casting and sugar-tong splinting. At the time of injury casts are usually split into two using a cast saw, known as bivalving, to allow for swelling and are overwrapped at a later time. By design sugar-tong splints allow for swelling and are overwrapped or converted to a cast at a later time. Traditionally long-arm casts have been used as the standard mode of immobilization for forearm fractures. Recent evidence demonstrates that long-arm casting is equivalent to better tolerated short-arm casting as an immobilization choice for distal third forearm fractures.1 Further work has shown that sugar-tong splints are also appropriate for treatment of distal third forearm fractures. No study has compared the efficacy of using a long-arm cast versus a sugar-tong splint for treatment of forearm shaft fractures.

ELIGIBILITY:
Inclusion Criteria:

* Single or both bone forearm shaft fractures, follow-up at the St. Louis Children's Hospital and affiliated branches

Exclusion Criteria:

* Children below 4 or above 12 years of age
* Distal radius/ulna fracture(s)
* Distal radius/ulna third shaft fracture(s)
* Proximal radius/ulna third shaft fracture(s)
* Radius/ulna fracture(s) not requiring reduction
* Open radius/ulna fracture(s)
* Radius/ulna fracture(s) requiring open reduction in the operating room
* Patient with metabolic defects
* Pathologic radius/ulna fracture(s)
* Previous fractures in the same location (radius/ulna)

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-03 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Radiographic measurements | 1 week
  Measure sagittal angulation
Radiographic measurements | 2 weeks
  Measure sagittal angulation
Radiographic measurements | 4 weeks
  Measure sagittal angulation
Radiographic measurements | 6 weeks
  Measure sagittal angulation
Radiographic measurements | 1 week
  Coronal angulation
Radiographic measurements | 2 weeks
  Coronal angulation
Radiographic measurements | 4 weeks
  Coronal angulation
Radiographic measurements | 6 weeks
  Coronal angulation
Radiographic measurements | 1 week
  Displacement
Radiographic measurements | 2 weeks
  Displacement
Radiographic measurements | 4 weeks
  Displacement
Radiographic measurements | 6 weeks
  Displacement
Radiographic measurements | 1 week
  Percent displacement
Radiographic measurements | 2 weeks
  Percent displacement
Radiographic measurements | 4 weeks
  Percent displacement
Radiographic measurements | 6 weeks
  Percent displacement

SECONDARY OUTCOMES:
Clinical follow-up | 1 week
  Treatment information
Clinical follow-up | 2 weeks
  Treatment information
Clinical follow-up | 4 weeks
  Treatment information
Clinical follow-up | 6 weeks
  Treatment information

CONTACTS AND LOCATIONS:
Locations (1):
- St. Louis Children's Hospital, St Louis, Missouri, United States

REFERENCES:
- [Background] Bohm ER, Bubbar V, Yong Hing K, Dzus A. Above and below-the-elbow plaster casts for distal forearm fractures in children. A randomized controlled trial. J Bone Joint Surg Am. 2006 Jan;88(1):1-8. doi: 10.2106/JBJS.E.00320. PMID 16391243
- [Background] Levy J, Ernat J, Song D, Cook JB, Judd D, Shaha S. Outcomes of long-arm casting versus double-sugar-tong splinting of acute pediatric distal forearm fractures. J Pediatr Orthop. 2015 Jan;35(1):11-7. doi: 10.1097/BPO.0000000000000196. PMID 24787302
- [Background] Kamat AS, Pierse N, Devane P, Mutimer J, Horne G. Redefining the cast index: the optimum technique to reduce redisplacement in pediatric distal forearm fractures. J Pediatr Orthop. 2012 Dec;32(8):787-91. doi: 10.1097/BPO.0b013e318272474d. PMID 23147621
- [Background] Alemdaroglu KB, Iltar S, Cimen O, Uysal M, Alagoz E, Atlihan D. Risk factors in redisplacement of distal radial fractures in children. J Bone Joint Surg Am. 2008 Jun;90(6):1224-30. doi: 10.2106/JBJS.G.00624. PMID 18519314